CLINICAL TRIAL: NCT03671642
Title: Perioperative Perfusion Measurement - a Feasibility and Usability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Nikolaj Albeck Nerup, PhD-fellow, senior resident, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: H-18006334
Record Dates: First submitted 2018-08-08; First posted 2018-09-14 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Esophageal Cancer
Keywords: perfusion; indocyanine green angiography; feasibility study
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perfusion assessment (Experimental): Q-ICG: quantitative perfusion assessment with FA White light perfusion assessment FA: fluorescence angiography without quantification
  Interventions: Device: Q-ICG; Procedure: White light perfusion assessment; Procedure: Fluorescence angiography

INTERVENTIONS:
Device: Q-ICG — Quantitative perfusion assessment with indocyanine green on a touch screen tablet
Procedure: White light perfusion assessment — Traditional visual perfusion assessment in white light
Procedure: Fluorescence angiography — Perfusion assessment with fluorescence angiography - without quantification

SUMMARY:
This study will investigate a new method to assess tissue perfusion during surgery for esophageal cancer.

When a tumor in the distal esophagus is removed, the ends of the esophagus and the stomach must be reconnected by an anastomosis. An optimal perfusion is essential to ensure a good healing of the anastomosis. If anastomotic leakage occurs, it may prolong hospital stay, increase the risk of serious complications and death, delay start-up of chemotherapy and worsen the long-term survival prognosis.

During the operation the blood supply to the ends of the esophagus and stomach will be assessed in different ways; The traditional where the surgeon looks and feels on the tissue, and newer methods with an indocyanine green and cameras that illuminate the tissue with near-infrared light. The surgeon will assess whether these methods change the decision on where the ends should be sewn together.

DETAILED DESCRIPTION:
Introduction:

An optimal perfusion is essential in gastrointestinal surgery when resection of a cancerous tissue requires an anastomosis, since impaired perfusion seems to be associated with increased risk of anastomotic leakage (AL). AL is a severe complication with the risk of; prolonged hospital stay, cancer recurrence, permanent stoma in colorectal surgery, and increased short and long-term mortality. To avoid poor perfusion of an anastomosis, perfusion assessment is necessary during the operative procedure. Traditionally, perfusion is assessed visually and manually by the surgeon by judging the; color of the tissue, bleeding from the resection line, and the arterial supply pulse by palpation. These methods have earlier been shown to be unreliable and prone to observer bias. Furthermore, palpation of arterial supply is not possible in laparoscopic or robot-assisted surgery, and the increased use of staplers to divide the bowel leaves no bleeding resection lines. Therefore newer methods for perfusion assessment have been investigated, and fluorescence angiography (FA) and laser speckle contrast imaging (LSCI) has shown very promising results. In a systematic review of nonrandomized studies, the leakage rate in 916 colorectal resections was significantly lower when using FA compared to controls (3.3%, [95% CI: 1.97-4.63%] vs 8.5%, [95% CI: 4.8-12.2%], p=0.0055).

In FA, the tissue of interest is exposed to near-infrared (NIR) light simultaneously with intravenous injection of a fluorescent dye. When the dye reaches the illuminated area, it fluoresces, and a camera with a special filter can visualize the microcirculation of the tissue on a monitor. Many NIR-camera systems are on the market, combining the technique with conventional laparoscopic or robotic equipment, and several non-randomized studies have indicated that FA may reduce the anastomotic leakage rate in gastrointestinal surgery. Most surgeons are using only a visual subjective assessment of the FA, which may be prone to observer bias. Moreover, if the camera is not held at a standard distance from the tissue, or a different concentration of dye is used, a false negative or positive assessment of the perfusion may be made. Therefore, it has been argued that there is a need for an objective unbiased quantitative assessment tool in FA.

A quantification algorithm that provides a fluorescence-time curve and a quantitative parameter of perfusion, the normalized slope has previously been published, where a nearly linear correlation to regional flow was found. Until now measurements has been performed as analyses of video-recordings after the procedure.

In order to use the method in a clinical setting, development and testing of a tool that may be operated by the surgeon during the procedure to perform perioperative measurements is of high importance. A touchscreen tablet has been developed, in order to perform live perioperative quantitative perfusion assessment using FA. The tool may be used with several systems including Karl Storz fluorescence laparoscopic equipment and the daVinci SI or XI from Intuitive. This tool is essential in order to implement the technology into daily practice, as it allows the surgeon to get an immediate quantitative parameter of perfusion (normalized slope) at desired regions of interest. The interface of the tool should be easy to use and provide fluorescence-time curves to control the automated calculation of the normalized slope. In addition, a color-coded map of perfusion intensity should be provided as an overlay on the white light picture of the bowel investigated.

Aim:

The touchscreen tablet has currently only been tested in animal surgery. The aim of the present study is to investigate if the use of a perioperative quantitative perfusion assessment tool may improve the perfusion assessment during surgery in humans.

Hypotheses:

* Perioperative perfusion assessment with FA will change the point of resection determined by conventional visual perfusion assessment in GI junctional procedures.
* Quantitative perfusion assessment with FA (Q-ICG) will further change the point of resection determined by visual assessment of the FA and conventional visual assessment of perfusion in GI junctional procedures.

Primary endpoints:

* Feasibility of perfusion assessment with traditional visual, visual FA, and Q-ICG - complied by completion rates.
* The feasibility and usability of the tool, the surgeons' experiences with the Q-ICG-tablet interface - rated on a validated questionnaire, the System Usability Scale.

Secondary endpoints:

• Differences in the distance from the determined resection points using traditional assessment, FA, and Q-ICG.

Methods

Study Design:

The study will be conducted as an observational feasibility and usability trial in patients undergoing open or robot-assisted resection of the gastroesophageal junction (GI junction) in a single university hospital center (Rigshospitalet, Department of Surgical Gastroenterology). Patients will serve as their own control. Demographic information (tumor-staging, gender, age, BMI, neoadjuvant treatment, ASA-classification, smoking, alcohol, medication etc.) will be collected from the electronic patient records. In addition, postoperative events, especially the presence of an anastomotic leakage, will be noted 30 days postoperatively. No formal sample size calculation has been performed as the study is a feasibility study. 20 patients will be included. Participating patients will receive the same standard post- and peri-operative care and follow-up as patients not included in the study.

Indocyanine green Indocyanine green (ICG) is a well-described nontoxic tricarbocyanine dye used for decades in ophthalmology, cardiology, and hepatology. Very few mild adverse reactions have been reported, but caution in patients with thyrotoxicosis, allergy towards iodine or indocyanine green should be made. When injected intravenously it binds to blood lipoproteins and is solely metabolized by the liver and excreted in the bile, with a short half-life of approximately 4-5 minutes.

Surgical procedure and perfusion assessment When the dissection and division of the feeding blood vessels are complete and the gastric conduit established and drawn to the thorax, the gastrointestinal surgeon will choose the most proximal point possible on the conduit for the anastomosis (Anastomotic point surgeon, APS) by pointing while a picture is captured, blinded for the thoracic surgeon. A sterile paper ruler will be introduced to the thorax, in order to measure the distance between the chosen resection points. Then, LSCI measurement of the conduit is performed, and finally, a bolus of ICG (0.25 mg/kg body weight) will be injected intravenously and flushed with 5 mL of saline, and the tissue of interest exposed to NIR-light (excitation wavelength 750-800 nm) and emission observed at 800 nm (FA). During the video-captures of LSCI and ICG-FA, the respiration will be paused for a maximum of 20 seconds initiated at the moment of saline injection. After the FA the thoracic surgeon will by visual assessment determine and mark a new anastomotic point by pointing at the most proximal point possible on the conduit for the anastomosis, while a picture is taken (anastomotic point fluorescence angiography, APFA). After the quantitative FA the surgeon will again mark an anastomotic point (APQFA). The final anastomotic point will be chosen by the primary gastrointestinal and the thoracic surgeon, and if the assessment of FA or quantitative FA will influence this decision is solely up to the surgeon. The same points will be marked on the LSCI picture but not revealed to the surgeon since the quantitative assessment of the LSCI demands on post hoc data-analysis.

When the surgeon decides how much tissue to resect to ensure an optimal anastomotic perfusion, care must be taken not to cause tension to the anastomosis by resecting too much of the gastric conduit or the esophagus, as tension is a known risk factor of anastomotic leakage. Again, the level of resection is solely decided by the surgeon and this decision should, as always, be made by balancing factors of tension, perfusion, and excessive tissue loss - all combined to ensure an optimal anastomotic healing.

Laparoscopic fluorescence angiography A laparoscope (ICG-Hopkins telescope 30°, 10 mm, Karl Storz Gmbh and Co. KG, Tüttlingen, Germany) will be connected to a camera system (IMAGE1, Karl Storz Gmbh and Co. KG, Tüttlingen, Germany) and a light-source (D-light P, Karl Storz Gmbh and Co. KG, Tüttlingen, Germany) will supply the excitatory light and record the FA. The laparoscope will be fixed in a mechanical holding arm 10 cm from the tissue of interest, ensuring a stable position throughout the experiment.

Robot-assisted fluorescence angiography A surgical robot DaVinci SI (Intuitive Surgical Inc., Sunnyvale, CA, USA) and the Firefly Fluorescence Imaging system will be used. The camera will be fixed 10 cm from the tissue of interest, ensuring a stable position throughout the experiment.

Quantitative fluorescence angiography (Q-ICG) A video capture device (Av.io HD™, Epiphan video, California, USA) will be connected to the surgical robot or the laparoscopic camera system and transfer the video capture to a tablet (Microsoft Surface Pro4 I5, Microsoft, Redmond, WA, USA). A program developed to quantify the FA will be installed. Here the operator can choose regions of interest to quantify from the captured video sequence. A color grading of perfusion will be provided as well as quantitative values from specific points. From this assessment, the surgeon will again determine a new resection point (APQFA).

Comparison of resection points The distance from the tumor to the RPS will be measured before the FA using the paper ruler. In addition, the distance from the APS to APFA and APQFA will be measured using the ruler, either during the procedure or post hoc using the video-capture. The comparison of the distance will be made on the distance of each point from the tumor.

Feasibility The feasibility will be investigated by comparison of completion rates of the different perfusion assessment methods; traditional, FA, Q-ICG.

Usability The usability of the quantitative perfusion assessment tool will be investigated with a validated questionnaire, the System Usability Scale, answered by the surgeon immediately after the procedure.

Statistics Comparison of data will be performed using Mann Whitney U test or a paired sample t-test depending on distribution normality. P-values < 0.05 is considered significant. No formal sample size calculation has been made, as the study is considered a feasibility trial. 20 patients will be recruited. Statistic evaluation was performed using IBM SPSS Statistics © (v 22.0 SPSS Inc. Chicago, IL, USA).

Adverse events, risks, and disadvantages Adverse events associated with the use of ICG are extremely rare and severe anaphylactic reactions are almost never occurring. However, safety precautions have been made by excluding patients with allergy to iodine, ICG or shellfish. In addition, no patients with liver insufficiency, thyrotoxicosis, ongoing pregnancy, or lactating women will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients (above 18 years) scheduled for planned open or robot-assisted resection of the gastroesophageal junction (GI junction) for GI junctional cancer.

Exclusion Criteria:

* Allergy towards; iodine, indocyanine green or shellfish
* Liver insufficiency
* Thyrotoxicosis
* Pregnancy or lactation
* Legally incompetent for any reason
* Withdrawal of inclusion consent at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Completion rates | during surgery
  Feasibility of perfusion assessment with traditional visual, visual FA, and Q-ICG

SECONDARY OUTCOMES:
Differences in resection points | up to 6 months
  Differences in the distance from the determined resection points using traditional assessment, LSCI, FA, and quantitative FA.
System Usability Scale | up to one week
  The feasibility and usability of the tool, the surgeons' experiences with the Q-ICG tablet interface - rated on a validated questionnaire, the System Usability Scale - https://www.usability.gov/how-to-and-tools/methods/system-usability-scale.html.
  Scores ranges from 0-100, where a score of 68 is considered average.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Achiam, MD,PhD,DMSci, Study Chair — Department of Surgical Gastroenterology, Rigshospitalet
Locations (1):
- Department of Surgical Gastroenterology - Rigshospitalet, Copenhagen Ø, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nerup N, Andersen HS, Ambrus R, Strandby RB, Svendsen MBS, Madsen MH, Svendsen LB, Achiam MP. Quantification of fluorescence angiography in a porcine model. Langenbecks Arch Surg. 2017 Jun;402(4):655-662. doi: 10.1007/s00423-016-1531-z. Epub 2016 Nov 15. PMID 27848028